CLINICAL TRIAL: NCT02485314
Title: Reliability and Validity of Turkish Version of the Participation and Environment Measure for Children and Youth
Brief Title: Reliability and Validity of Turkish Version of PEM-CY
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ozgun Kaya Kara, PT, PhD, Assist. Prof, Hacettepe University
Other Study IDs: GO14/553
Record Dates: First submitted 2015-06-10; First posted 2015-06-30 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Child
Keywords: children; disability; family; participation

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participation: Parents will complete the PEM-CY (Participation and Environment Measure for Children and Youth).
  Interventions: Other: Participation

INTERVENTIONS:
Other: Participation — The PEM-CY will be field-tested with a sample of 650 caregivers of children with and without disabilities residing in the Turkey.
  Other Names: PEM-CY

SUMMARY:
The Participation and Environment Measure for Children and Youth (PEM-CY) is the first instrument that combines parental assessment of children's participation in home, school, and community activities with qualities of each environment that are perceived to support or hinder participation. This combined format may help to clarify the relative impact of environmental factors (including the natural and built environment), compared to personal factors, on children's participation in specific settings. The aim of this study was to examine reliability and validity of Turkish version of the Participation and Environment Measure for Children and Youth (PEM-CY).

DETAILED DESCRIPTION:
The International Classification of Functioning, Disability and Health-Child and Youth Version (ICF-CY; WHO 2007) is designed to guide assessment and intervention efforts to minimize disparities in children's participation. Participation is defined in the ICF-CY as ''involvement in life situations'' and is further conceptualized as a multidimensional construct with both objective (e.g., frequency) and subjective (e.g., satisfaction) dimensions. Participation is linked to contextual factors, including: 1) personal factors (child personal factors such as child's age, gender, and functional abilities; family demographic factors); and 2) features of environments (physical (natural and built), social, attitudinal, and institutional factors, and availability and adequacy of resources). Since its adoption in the ICF-CY, an increasing number of participation measures have been developed. Among these measures, the Participation and Environment Measure for Children and Youth (PEM-CY) is the first instrument that combines parental assessment of children's participation in home, school, and community activities with qualities of each environment that are perceived to support or hinder participation. This combined format may help to clarify the relative impact of environmental factors (including the natural and built environment), compared to personal factors, on children's participation in specific settings.

ELIGIBILITY:
Inclusion Criteria:

* they will identify themselves as a parent or legal guardian of the child who is the focus of the study
* they are able to read Turkish
* their child is between 5 and 17 years old at the time of enrolment.

Exclusion Criteria:

* who don't want to attend the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Caregivers of children with and without disabilities
Sampling Method: Probability Sample
Enrollment: 470 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Participation and Environment Measure for Children and Youth with and without disability as a measure of participation | 1 year
  The PEM-CY will be applied for once for 500 participants. • A comparison will be made between results of children with disabilities and healthy children to test the validity of the Turkish version of PEM-CY.

SECONDARY OUTCOMES:
Variation in participation and environment measure for children and youth with and without disability | 1 year
  Investigate the intraclass correlation coefficient of Turkish version of PEM-CY was used to calculate test retest reliability. PEM-CY was administered twice within a period of 1 week to participants in order to test the test-retest reliability of the scale.
Correlation between different items of Participation and Environment Measure for Children and Youth with and without disability | 1 year
  Investigate the internal consistency reliability of Turkish version of PEM-CY by using Cronbach's alpha coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Ozgun Kaya Kara, PhD, Study Director — Akdeniz University; Duygu Turker, PhD, Principal Investigator — Saglik Bilimleri Universitesi Gulhane Tip Fakultesi; Koray Kara, Assist. Prof, Principal Investigator — Antalya Training and Research Hospital
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khetani MA, Cliff AB, Schelly C, Daunhauer L, Anaby D. Decisional Support Algorithm for Collaborative Care Planning using the Participation and Environment Measure for Children and Youth (PEM-CY): A Mixed Methods Study. Phys Occup Ther Pediatr. 2014 Mar 26. doi: 10.3109/01942638.2014.899288. Online ahead of print. PMID 24670061
- [Background] Coster W, Bedell G, Law M, Khetani MA, Teplicky R, Liljenquist K, Gleason K, Kao YC. Psychometric evaluation of the Participation and Environment Measure for Children and Youth. Dev Med Child Neurol. 2011 Nov;53(11):1030-7. doi: 10.1111/j.1469-8749.2011.04094.x. PMID 22014322
- [Background] Coster W, Law M, Bedell G, Liljenquist K, Kao YC, Khetani M, Teplicky R. School participation, supports and barriers of students with and without disabilities. Child Care Health Dev. 2013 Jul;39(4):535-43. doi: 10.1111/cch.12046. PMID 23763254
- [Background] Chien CW, Rodger S, Copley J, Skorka K. Comparative content review of children's participation measures using the International Classification of Functioning, Disability and Health-Children and Youth. Arch Phys Med Rehabil. 2014 Jan;95(1):141-52. doi: 10.1016/j.apmr.2013.06.027. Epub 2013 Jul 12. PMID 23851418